CLINICAL TRIAL: NCT06248528
Title: To Compare the Survival Differences in Patients With HCC and Portal Vein Tumor Thrombosis Treated With Liver Resection-based Therapy Versus Locoregional-based Therapy: a Prospective Cohort Study
Brief Title: Comparing the Prognosis of Patients With HCC and PVTT Treated With Surgery Versus Locoregional Therapy.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma; Adjuvant therapy; Overall survival; Liver resection; Combined therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liver resection-based group (Experimental): Patients in the liver resection-based group received adjuvant PD-1 inhibitors plus targeted drugs following liver resection.
  Interventions: Procedure: Liver resection
- Locoregional treatment-based group (Active Comparator): Patients in the locoregional treatment-based group received PD-1 inhibitors plus targeted drugs following locoregional therapy.
  Interventions: Procedure: Locoregional therapy

INTERVENTIONS:
Procedure: Liver resection — Patients in the intervention group received liver resection and postoperative adjuvant therapy
  Arms: Liver resection-based group
Procedure: Locoregional therapy — Patients in the control group received locoregional therapy and systemic therapy
  Arms: Locoregional treatment-based group

SUMMARY:
Hepatocellular carcinoma is prone to invade the portal vein and form portal vein thrombosis, and patients in this period are directly included in the advanced stages, i.e. Barcelona clinical liver cancer stage C. For the treatment of PVTT, there are differences between Eastern and Western guidelines, with systemic drugs being the standard of care in Western countries, while surgical treatment is often actively practiced in the Asia-Pacific region. More research is needed to explore the differences between these two approaches.

DETAILED DESCRIPTION:
Hepatocellular carcinoma is prone to invade the portal vein and form portal vein thrombosis, and patients in this period are directly included in the advanced stages, i.e. Barcelona clinical liver cancer stage C. For the treatment of PVTT, there are differences between Eastern and Western guidelines, with systemic drugs being the standard of care in Western countries, while surgical treatment is often actively practiced in the Asia-Pacific region. In recent years, breakthroughs have been made in the treatment of advanced HCC, and systemic drug combinations such as PD-1 inhibitors combined with targeted therapies, and local area therapy combined with systemic therapy have shown excellent anti-tumor effects. Postoperative adjuvant therapy is also advancing, and the combination of adjuvant systemic medications for patients after PVTT has also been effective in reducing postoperative recurrence. Which approach is better for PVTT patients needs to be explored in depth.

We launched the CHALLENGE-01 study in October 2023. The study consists of two phases: the first phase involves retrospective data collection from 2019 to 2023 and prospective follow-up of survival information. Specifically, the liver resection+ PD-1 inhibitor + lenvatinib (LRPL) cohort included 225 cases, the TACE + PD-1 inhibitor + lenvatinib (TPL) cohort included 205 cases, and the surgery-only treatment cohort included 200 cases as an additional control group. Data analysis from the first phase of the study showed that the median follow-up times for the LRPL and TPL cohorts were 31.6 months and 22.5 months, respectively. Based on retrospective cohort data, we calculated the sample size required for the prospective study (446) and formally initiated the second-phase prospective clinical trial in January 2024. The study completed the required enrollment from nine centers in China by December 31, 2024, but has not yet reached the primary endpoint (OS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years
* Pathological type is HCC, and with PVTT
* No extrahepatic HCC
* Eastern Cooperative Oncology Group (ECOG) performing status of 0-1 and Child-Pugh grade A for the liver resection group
* ECOG performing status of 0-2 and Child-Pugh grade A-B for the locoregional-based group
* Adequate hematologic and organ function

Exclusion Criteria:

* Any history of other malignant tumors or recurrent HCC
* Any acute active infectious diseases, active or history of autoimmune disease, or immune deficiency
* Any persistent serious liver resection or locoregional therapy-related complications
* Esophageal and/or gastric variceal bleeding within 6 months
* Inability or refusal to comply with the treatment and monitoring
* Participation in other clinical trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1076 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of include in this research until the date of death from any cause, whichever came first, assessed up to 60 months.
  Overall survival was defined as the period from study inclusion until death from any cause.

SECONDARY OUTCOMES:
Adverse effects | 12 months
  Adverse reactions are defined as any reaction during treatment that is inconsistent with the purpose of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: WanGuang Zhang, Study Director — Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No